CLINICAL TRIAL: NCT06861634
Title: Optimization of Morphinomimetic Administration Intraoperatively: Evaluation of the Impact of the NOL Index on the Occurrence of Postoperative Adverse Events Related to Morphinomimetics: A Randomized Controlled Trial
Brief Title: Optimization of Morphinomimetic Administration Intraoperatively: Evaluation of the Impact of the NOL Index on the Occurrence of Postoperative Adverse Events Related to Morphinomimetics
Acronym: NOL-Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DR220248
Record Dates: First submitted 2025-02-13; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia; Intensive Care Medicine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group NOL (Experimental): Morphinomimetics will be administered according to NOL Index values.
  Interventions: Procedure: Nol index
- Group control (No Intervention): Morphinomimetics will be administered according to the usual criteria.

INTERVENTIONS:
Procedure: Nol index — Morphinomimetics will be administered according to NOL Index values or according to the usual criteria.
  Arms: Group NOL

SUMMARY:
Reducing the quantity of morphinomimetics during the operative period reduces the prevalence and intensity of adverse effects.

However, morphinomimetics are indispensable during surgery, as they limit the autonomic nervous system's deleterious reactions to nociception. The administration of these drugs in intravenous boluses during surgery is usually guided by their duration of action and by variations in heart rate and blood pressure. Other events, such as hypovolemia or extreme surgical position, may stimulate the autonomic nervous system outside of nociception. These events, along with routine drug administration, can lead to undue consumption of morphinomimetics.

The Nol index, a multiparametric monitor of nociception, is based on analysis of variations in plethysmography waveform, heart rate and skin conductance. It has been demonstrated that the use of this type of monitor can reduce intraoperative consumption of morphinomimetics and optimize their administration. Does intraoperative morphinomimetic administration optimized by the NOL index have an impact on the occurrence of dose-dependent adverse effects?

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Subject aged ≥ 18 years
* Affiliated with a social security scheme
* Having given written informed consent to participate study
* Admitted for major surgery expected to last more than 2 hours
* Under general anesthesia with tracheal intubation
* For a planned hospital stay of at least 48 hours
* Participant's ability to understand the nature and objectives of the study to comply with study requirements.

Exclusion Criteria:

* Contraindication to one of the drugs used for anesthesia
* Urgent surgery
* Intracranial surgery
* Transplant surgery
* Cardiac surgery
* Surgery with scheduled local anesthesia
* Patient requiring postoperative intubation
* Neuromuscular disease
* Patient chronically using morphinomimetics
* Chronic pain patient
* Patients with a history of sleep apnea
* Conditions likely to interfere with photoplethysmograph signal acquisition or skin conductance (excessive or tremors of the extremities, skin lesions or burns)
* Patients wearing false nails and/or nail polish
* Contraindication to the use of the PMD 200 ™ medical device (including cardiovascular resuscitation and cardioversion/defibrillation);
* Patient with an implanted pacemaker or defibrillator
* Treatment with β-blockers
* Preoperative cardiac arrhythmia
* Pregnant or breast-feeding women. A β-HCG test will be systematically performed prior to inclusion of non-menopausal women menopausal women
* Patients under legal protection (safeguard of justice, curatorship guardianship) or deprived of liberty
* Participation in other interventional research involving an experimental drug or medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Composite outcome including at least one occurrence of hypoxemia, of nausea-vomiting or of ileus. | From enrollment to within 48 hours post-extubation.
  1. occurrence of hypoxemia: at least 1 episode of SpO2 < 95%,
  2. occurrence of nausea-vomiting: at least one episode of nausea requiring antiemetic treatment, or at least one episode of vomiting,
  3. occurrence of ileus: absence of gas or stool.

SECONDARY OUTCOMES:
Total consumption of intraoperative morphinomimetics | From intervention to 48 hours after extubation
Total consumption of intraoperative vasoconstrictors | From induction to extubation, up to 8 hours
  type of vasoconstrictor, amount of vasaoconstrictor used and number of boli of vasoconstrictor will be considered
Time of extubation | From the end of anesthesia administration to extubation, up to 1 hours
  Delay between the end of the hypnotic infusion and the patient becoming conscious and able to breathe freely
Time from extubation to theoretical post-anesthesia care unit discharge time with Aldrete score at 10 | From extubation to Aldrete score at 10, every 5 minutes, up to 2 hours
  Aldrete's score will be assessed every 5 minutes during his stay in the post-anesthesia care unit. Discharge from the post-anesthesia care unit will be possible when the Aldrete score reaches 10.
Maximum intensity of pain | From extubation to 48 hours postoperative
  Numeric rating scale (NRS): Patients rate their pain intensity on a 11-point Numeric Rating Scale (NRS-11), where 0 indicates the absence of pain and 10 means the worst possible pain.
Number of episodes of pain | From extubation to 48 hours postoperative.
  Numerical scale > 3
Number of episodes of hypoxemia | From intervention to 48 hours post-extubation
Number of episodes of nausea and vomiting | From intervention to 48 hours post-extubation
Hospital stay length | From admission to hospital discharge up to 1 month.
  Time from hospital admission to hospital discharge
Quality of post-operative recovery | From enrollment to 24 hours and 48 hours after chirurgical intervention
  The French version of the Quality of Recovery -15 (FQoR-15) is is a validated multidimensional PROM-based questionnaire that measures postoperative quality of recovery. The QoR-15 scale consists of 15 questions, where the patient is asked to quote dimensions of his/her recovery from 0 to 10. After summing all 15 responses, the QoR-15 is presented as a score, ranging from 0 to 150, with 150 corresponding to an ideal health status.
Intensity of chronic pain | At 3 months, at 6 months and at 12 months (end of the study)
  Phone contact : DN4 form The DN4 form (douleur neuropathique - neuropathic pain 4) is a form with 10 questions. The results are from 0 to 10. A result greater than 4 is considered positive.
Occurrence of hypoxemia | From enrollment to 48 hours post-extubation
  Occurrence of hypoxemia: at least 1 episode of SpO2 < 95%
Occurrence of nausea-vomiting | From enrollment to 48 hours post-extubation
  Occurrence of nausea-vomiting: at least one episode of nausea requiring antiemetictreatment, or at least one episode of vomiting
Occurrence of ileus | From enrollment to 48 hours post-extubation
  Occurrence of ileus: absence of gas or stool.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Chu Angers, Angers
  - CH BLOIS, Blois
  - Chu Brest, Brest
  - Chu Nantes, Nantes
  - Chru Tours Sar1, Tours
  - Chru Tours Sar2, Tours

IPD SHARING:
Plan to Share IPD: No